CLINICAL TRIAL: NCT02554955
Title: Pilot, Single-arm, Non-comparative, Open-label Study of Daclizumab in Combination With Mycophenolate Mofetil and Sirolimus in the Prevention of Acute Rejection in Cardiac Allografts Recipients in Risk of Deteriorated Renal Function
Brief Title: A Study of Daclizumab (Zenapax) in Combination With Mycophenolate Mofetil (CellCept) and Sirolimus in Prevention of Acute Rejection in Heart Transplant Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17910
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Daclizumab; Mycophenolic Acid

ARMS (1):
- Daclizumab + Mycophenolate mofetil (Experimental): Participants will receive intravenous (IV) daclizumab (2 milligrams per kilogram [mg/kg] within 6 hours after transplantation and 1 mg/kg every 2 weeks for a total of five doses), along with mycophenolate mofetil (one dose of 1.5 mg within 12 hours pretransplant, 1.5 mg twice daily [BID] within first week and 1 grams per day [g/day] BID from second week onwards) and sirolimus (3 mg/day) for 6 months.
  Interventions: Drug: Daclizumab; Drug: Mycophenolate mofetil; Drug: Silrolimus

INTERVENTIONS:
Drug: Daclizumab — Participants will receive IV daclizumab (2 mg/kg within 6 hours after transplantation and 1 mg/kg every 2 weeks) for a total of five doses.
  Other Names: Zenapax
Drug: Mycophenolate mofetil — Participants will receive mycophenolate mofetil orally (one dose of 1.5 mg within 12 hours pretransplant, 1.5 mg BID within first week and 1 g/day BID from second week onwards) for 6 months.
  Other Names: CellCept
Drug: Silrolimus — Participants will receive sirolimus orally (3 mg/day) for 6 months.

SUMMARY:
This study will evaluate the efficacy and safety of intravenous daclizumab in combination with oral mycophenolate mofetil and oral sirolimus in participants receiving a heart transplant, and at risk of impaired kidney function. The anticipated time on study treatment is 6 months, and the target sample size is 44 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than 18 years of age
* Single organ (heart) transplant recipients
* At risk for post-transplant renal dysfunction

Exclusion Criteria:

* Previous organ transplant
* Previous treatment with mycophenolate mofetil, daclizumab or sirolimus
* Positive for human immunodeficiency virus (HIV) infection
* History of malignancy within the last 5 years, except localized and treated skin cancer, treated and without evident relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with reported biopsy proven acute rejection episodes | up to 6 months

SECONDARY OUTCOMES:
Incidence of adverse events | up to 6 months
Incidence of Opportunistic Infections | Up to 5 years post transplant
Patient and graft survival | up to 6 months
Number of participants with malignancies | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (11):
- Spain (11):
  - A Coruña
  - Barcelona
  - El Palmar Murcia
  - L'Hospitalet de Llobregat
  - Madrid
  - Oviedo
  - Pamplona
  - Santander
  - Seville
  - Valencia
  - Valladolid